CLINICAL TRIAL: NCT04112758
Title: The Effect of Long-term High-intensity Interval Training on Conflict Monitoring in Children With ADHD: an ERP and sLORETA Study
Brief Title: Exercise Intervention on Conflict Monitoring in Children With Attention-deficit Hyperactivity Disorder
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Jung Tsai, Doctoral student, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201903HM013
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Exercise Intervention
Keywords: HIIT; executive function; ADHD; chronic exercise
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The group will receive twice a week for 5 week
  Interventions: Other: High-intensity interval training
- Control group (No Intervention): The group will be maintained their normal after school activities

INTERVENTIONS:
Other: High-intensity interval training — 2 times weekly for 5 weeks Circuit training with 4 stations
  Arms: Exercise group

SUMMARY:
The study mainly investigates the effect of high-intensity interval training on conflict monitoring in children with ADHD by using event-related potential and sLORETA techniques.

DETAILED DESCRIPTION:
The present study will have two experiments, one is a cross-section study and the other is intervention study.

As for cross-section study, typical developmental children and children with ADHD will perform the stroop task while recording their brain waves.

The intervention is twice a week for 5 weeks and before and after the intervention, children with ADHD will randomly assign to either an exercise group or control group. They will perform the stroop task while recording their brain waves.

ELIGIBILITY:
Inclusion Criteria:

1. age between 7 and 12 years
2. diagnosed with ADHD by a pediatric psychiatrist, which is not required for TD
3. no history of brain injury or neurological conditions, such as exhibited epileptic seizures, serious head injuries, and periods of unconsciousness.

Exclusion Criteria:

1. cannot follow the instruction
2. cannot complete all the procedure

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-01-23 (Actual)

PRIMARY OUTCOMES:
Behavioral performance | Day 0 and post-intervention at Week 5
  reaction time (ms) is generated by computerized task deﬁned as correct responses within the range from 200-1500 ms
Behavioral performance | Day 0 and post-intervention at Week 5
  response accuracy (percentage) is generated by computerized task defined as percentage of trials that successfully responded to target stimulus

SECONDARY OUTCOMES:
N2 & P3 components | Day 0 and post-intervention at Week 5
  Electroencephalographic (EEG) activity will be measured at 64 sites. The amplitude of the N2 is deﬁned as the mean amplitude within a 50-ms interval surrounding the maximal negative peak within a 200- to 400-ms latency window.
  The amplitude of the P3 is deﬁned as the mean amplitude within a 50-ms interval surrounding the maximal positive peak within a 300- to 800-ms latency window.

OTHER OUTCOMES:
Brain activation | Day 0 and post-intervention at Week 5
  To examine sources relating to amplitude in ERPs, source localization will be conducted using standardized low resolution brain electromagnetic tomography (sLORETA) The sLORETA analysis with the ERP data will be selected by four 100 ms bins covering the period from 0 to 200 ms after stimulus-onset (0-50, 50-100, 100-150, and 150-200 ms).

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No